CLINICAL TRIAL: NCT04435821
Title: Use of PET/MRI in the Diagnosis of Pediatric Chronic Pain
Brief Title: PET/MRI in the Diagnosis of Pediatric Chronic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Helen Ruth Nadel, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 52830
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Pediatric Disorder; Neuropathic Pain; Nociceptive Pain
Keywords: PET/MRI; Pediatric Chronic Pain
MeSH Terms: conditions — Chronic Pain; Neuralgia; Nociceptive Pain | interventions — 6-(3-fluoropropyl)-3-(2-(azepan-1-yl)ethyl)benzo(d)thiazol-2(3H)-one

STUDY DESIGN:
Intervention Model Description: Pediatric Chronic Pain Patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pediatric Chronic Pain Patients (Experimental): Individuals 11-18 years old, with chronic pain (lasting at least 2 months).
  Interventions: Drug: [18F]FTC-146

INTERVENTIONS:
Drug: [18F]FTC-146 — Participants will be injected with 0.08 mCi/kg [18F]FTC-146. A whole-body PET/MRI scan will be performed after injection.
  Other Names: S1R

SUMMARY:
[18F]FTC-146 is a sigma-1 receptor detector and is an experimental radiotracer. Several studies have implicated involvement of sigma-1 receptors in generation and perpetuation of chronic pain conditions, while others are investigating anti sigma-1 receptor drugs for treatment of chronic pain. Using [18F]-FTC-146 and PET/MRI, we hope to learn what is the best approach to identify the source of pain generation and characterize the disease in pediatric patients with chronic pain.

DETAILED DESCRIPTION:
It is estimated that 20% to 35% of children and adolescents worldwide are affected by chronic pain. As a result of chronic pain, children may miss school, withdraw from social activities, and develop internalizing behaviors. Therefore, accurately identifying the cause of a child's pain is important for both proper treatment of the pain and to prevent problems secondary to the chronic pain. Evidence in the literature points strongly toward an involvement of the sigma-1 receptor in neurogenic inflammation, which is known to be an important pathophysiological mechanism for maintenance and perpetuation of chronic neuropathic pain. The investigators hope to image and identify activated pain pathways in pediatric pain paitents using a radiolabeled biomarker for increased S1R expression. By localizing and quantifying areas of increased S1R expression to sites of augmented nociceptive activity using hybrid molecular/anatomic imaging techniques, we will objectively identify sites of neurogenic inflammatory activity and pain generation. The ability to image the changes associated with chronic pain generating pathologies provides us with a tool to identify and measure the intensity of the pathology. Imaging S1R expression in chronic pain states in pediatric patients would be both novel in its application and extremely powerful in better characterizing pediatric pain.

ELIGIBILITY:
Inclusion Criteria:

* 11-18 years old.
* Chronic pain (nociceptive, neuropathic or mixed pain) lasting at least 2 months.
* Pain level of at least 4/10 on a 0-10 Comparative Pain Scale (reported at time of screening).
* Covid Vaccination status: Vaccinated or unvaccinated subjects who received a negative test result from the Covid test within 72 hours of the scan.

Exclusion Criteria:

* MRI incompatible
* Pregnant or nursing
* Non-English speaker
* Claustrophobic

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
[18F]FTC-146 Biodistribution in Pain Patients [18F]FTC-146 Biodistribution in Pain Patients [18F]FTC-146 Biodistribution in Pain Patients | 3 hours
  Biodistribution of [18F]FTC-146 represented as Standardized Uptake Value max (SUVmax) in pain patients.

CONTACTS AND LOCATIONS:
Overall Officials: Helen R Nadel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No